CLINICAL TRIAL: NCT06231290
Title: The Influence of Magnification and Clinical Experience on the Outcome of Pulpotomy in Mature Adult Teeth: A Randomized Clinical Trial
Brief Title: The Influence of Magnification and Clinical Experience on the Outcome of Pulpotomy in Mature Adult Teeth
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Mohamed Ahmed Mohamed Yahia, Postgraduate student, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 874/3036
Record Dates: First submitted 2024-01-20; First posted 2024-01-30 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Irreversible Pulpitis
Keywords: Pulpotomy; Magnification; Clinical experience; Irreversible pulpitis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Postgraduate operator with magnification (Active Comparator)
  Interventions: Other: Adult full pulpotomy procedure
- Postgraduate operator without magnification (Experimental)
  Interventions: Other: Adult full pulpotomy procedure
- Undergraduate operator with magnification (Experimental)
  Interventions: Other: Adult full pulpotomy procedure
- Undergraduate operator without magnification (Experimental)
  Interventions: Other: Adult full pulpotomy procedure

INTERVENTIONS:
Other: Adult full pulpotomy procedure — The adult pulpotomy procedure of mature molars will be carried out with the use of magnification (dental loupes or microscope) in healthy patients. The procedure will be performed either by postgraduate or undergraduate operators.

SUMMARY:
The goal of this interventional randomized clinical trial is to test the effect of magnification and clinical experience of the operator on the success rate of full pulpotomy in mature adult molar teeth.

The main questions it aims to answer are:

* Does the use of magnification raise the success rate of full pulpotomy of mature adult molars?
* Does the clinical experience of the operator dentist raise the success rate of full pulpotomy of mature adult molars?

Participants will be asked to do the following:

* Receive the pulpotomy treatment of their target molar tooth.
* Record the pain score in the pain assessment chart.
* Attend the follow-up visits. They'll receive a full pulpotomy treatment of their target molar tooth. Researchers will evaluate the usage of magnification in performing the pulpotomy procedure of adult molar teeth by postgraduate or undergraduate operators in comparison to performing the same pulpotomy procedure without magnification to see if it raises the overall success rate of pulpotomy.

ELIGIBILITY:
Inclusion Criteria:

* Healthy patients diagnosed with acute irreversible pulpitis related to maxillary or mandibular permanent molar teeth without apical periodontitis.

Exclusion Criteria:

* Non-vital teeth.
* Immature teeth.
* Presence of swelling or sinus tract.
* Teeth with mobility grade II or III.
* Immunocompromised patients.
* Non-restorable teeth.
* Teeth with apical periodontitis seen in periapical radiograph.
* Periodontally affected teeth.
* Teeth with reversible pulpitis
* Extensive non-stoppable bleeding more than 6 minutes
* Teeth with partial necrosis

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Estimated)
Dates: Start 2024-03-20 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Clinical and radiographic outcome | Immediately, 1, 3, 6 and 12 months.
  The clinical outcome will be measured by the presence or absence of signs and symptoms. The radiographic outcome will be measured by using the PAI index which is a scale from 1 (best) to 5 (worst).

SECONDARY OUTCOMES:
Postoperative pain | Immediately, 24, 48, 72 hours and 7 days
  The postoperative pain will be measured by the modified Verbal Descriptor Scale which is a scale from 0 (best) to 10 (worst).

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dental Medicine, Al-Azhar University, Cairo, Egypt